CLINICAL TRIAL: NCT04609969
Title: Diagnostic Performance Evaluation of a Novel SARS-CoV-2 (COVID-19) Antigen Detection Test on Nasopharyngeal Specimens i
Brief Title: Diagnostic Performance Evaluation of a Novel SARS-CoV-2 (COVID-19) Antigen Detection Test
Acronym: COVID-VIRO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHRO-2020-18
Record Dates: First submitted 2020-10-28; First posted 2020-10-30 (Actual); Last update posted 2020-12-07 (Actual); Status verified 2020-12

CONDITIONS: Covid19; SARS-CoV-2 Infection
Keywords: SARS-CoV-2 infection; COVID19; Antigen detection test
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Two concurrent nasopharyngeal swab specimens are collected for each participant. Comparison between RT-qPCR and COVID-VIRO® results of RT-qPCR positive patients is used to assess COVID-VIRO® sensitivity. Conversely, comparison between RT-qPCR and COVID-VIRO® results of RT-qPCR negative patients is used to assess COVID-VIRO® specificity.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Comparison between RT-qPCR and COVID-VIRO® results on nasopharyngeal swab specimens (Experimental): Two concurrent nasopharyngeal swab specimens are collected for each participant. Comparison between RT-qPCR and COVID-VIRO® results of RT-qPCR positive patients is used to assess COVID-VIRO® sensitivity. Conversely, comparison between RT-qPCR and COVID-VIRO® results of RT-qPCR negative patients is used to assess COVID-VIRO® specificity.
  Interventions: Diagnostic Test: RT-qPCR test; Diagnostic Test: COVID-VIRO® test

INTERVENTIONS:
Diagnostic Test: RT-qPCR test — Two concurrent nasopharyngeal swab specimens are collected for each participant. Comparison between RT-qPCR and COVID-VIRO® results of RT-qPCR positive patients is used to assess COVID-VIRO® sensitivity. Conversely, comparison between RT-qPCR and COVID-VIRO® results of RT-qPCR negative patients is used to assess COVID-VIRO® specificity.
Diagnostic Test: COVID-VIRO® test — Two concurrent nasopharyngeal swab specimens are collected for each participant. Comparison between RT-qPCR and COVID-VIRO® results of RT-qPCR positive patients is used to assess COVID-VIRO® sensitivity. Conversely, comparison between RT-qPCR and COVID-VIRO® results of RT-qPCR negative patients is used to assess COVID-VIRO® specificity.

SUMMARY:
The current prospective study was designed to assess the diagnostic specificity and sensitivity of a novel antigen-based rapid detection test (COVID-VIRO®) on nasopharyngeal specimens in comparison to the reference test in a real-life setting

DETAILED DESCRIPTION:
Two nasopharyngeal swab specimens will be concurrently collected on:

* adult patients hospitalized in the Infectious Diseases Department of the Centre Hospitalier Régional d'Orléans (CHRO) for confirmed SARS-CoV-2 infection,
* or symptomatic or asymptomatic subjects voluntarily accessing the COVID-19 Screening Department of the CHRO to perform a diagnostic test. COVID VIRO® diagnostic.

Specificity and sensitivity are assessed in comparison to real-time RT-qPCR results.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18 years old) already having a SARS-CoV-2 RT-qPCR positive result within 5 days
* Adult patients (>18 years old) requiring a SARS-CoV-2 RT-qPCR on nasopharyngeal swab specimen for any reason

Exclusion Criteria:

* Patients non wishing to participate
* Under guardianship or curatorship or safeguard of justice patients
* Inability to join the hospital other than by public transport

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2020-10-13 (Actual); Primary Completion 2020-10-17 (Actual); Study Completion 2020-10-17 (Actual)

PRIMARY OUTCOMES:
Evaluation of COVID VIRO® diagnostic specificity | Month 1
  COVID-VIRO® specificity is calculated using the RT-qPCR results as reference test, according to the following formulas:
  Specificity (%) = 100 x [Negative / (Negative + Positive)]
Evaluation of COVID VIRO® diagnostic sensitivity | Month 1
  COVID-VIRO® sensitivity is calculated using the RT-qPCR results as reference test, according to the following formulas:
  Sensitivity (%) = 100 x [Positive/ (Positive + Negative)]

SECONDARY OUTCOMES:
Evaluation of COVID VIRO® diagnostic sensitivity for RT-qPCR Cycle threshold value < or > 28 | Month 1
  COVID-VIRO® sensitivity is calculated using the RT-qPCR results, restricting for Cycle threshold value

CONTACTS AND LOCATIONS:
Overall Officials: Thierry PRAZUCK, Dr, Principal Investigator — CHR ORLEANS
Locations (1):
- Centre Hospitalier Régional d'Orléans, France, Orléans, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Drame M, Tabue Teguo M, Proye E, Hequet F, Hentzien M, Kanagaratnam L, Godaert L. Should RT-PCR be considered a gold standard in the diagnosis of COVID-19? J Med Virol. 2020 Nov;92(11):2312-2313. doi: 10.1002/jmv.25996. Epub 2020 Jul 14. No abstract available. PMID 32383182
- [Background] Zitek T. The Appropriate Use of Testing for COVID-19. West J Emerg Med. 2020 Apr 13;21(3):470-472. doi: 10.5811/westjem.2020.4.47370. PMID 32302278
- See also: WHO coronavirus Dashboard on Sept 15th,2020 — https://covid19.who.int/
- See also: France Epidemiologic situation on 2020 september 20th — https://www.santepubliquefrance.fr/dossiers/coronavirus-covid-19